CLINICAL TRIAL: NCT01544205
Title: fMRI Based Neurofeedback as a Treatment Method for Depression
Brief Title: Neurofeedback as a Treatment Tool for Depression
Acronym: NFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: Medical Research Council (Other Government); National Institute for Social Care and Health Research (Unknown)
Responsible Party: Principal Investigator, David Linden, Professor of Translational Neuroscience, Cardiff University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPON927-11; G 1100629 (Other Grant/Funding Number: MRC); HS/10/25 (Other Grant/Funding Number: NISCHR); 11/WA/0106 (Other: NHS Research Ethics Committee)
Record Dates: First submitted 2012-02-23; First posted 2012-03-05 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Unipolar Depression
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Emotion network up-regulation (Experimental): Participants use fMRI-based neurofeedback to train the upregulation of brain areas that respond to positive affective pictures (as identified during a functional localiser scan).
  Interventions: Other: fMRI-based neurofeedback
- Place processing network up-regulation (Active Comparator): Participants use fMRI-based neurofeedback to train the upregulation of brain areas that respond to place and house pictures (as identified during a functional localiser scan).
  Interventions: Other: fMRI-based neurofeedback

INTERVENTIONS:
Other: fMRI-based neurofeedback — 5 sessions lasting one hour each

SUMMARY:
The purpose of the study is to investigate whether neurofeedback delivered via functional magnetic resonance imaging signals can be used to train depressed patients to self-regulate emotion networks and whether this improves clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* major depressive disorder (MDD) diagnosis
* stable antidepressant dose medication

Exclusion Criteria:

* Other physical or psychiatric disorders
* Current substance abuse
* Current psychotherapy or other specific intervention
* Exclusion criteria applicable to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hamilton Depression Rating Scale (HDRS) score at the end of intervention (after 5th session) | Before start trial (baseline), after intervention (appr. 2 months)

SECONDARY OUTCOMES:
Change from Baseline in Hamilton Depression Rating Scale (HDRS) score at follow-up | Baseline, 3-month follow-up
Change from Baseline in Hospital Anxiety and Depression Scale (HADS) anxiety score at the end of intervention (after 5th session) | Baseline, end of intervention (appr. 2 months)
Change from Baseline in Hospital Anxiety and Depression Scale (HADS) anxiety score at follow-up | Baseline, 3-month follow-up
Change from Baseline in Hospital Anxiety and Depression Scale (HADS) depression score at the end of intervention (after 5th session) | Baseline, end of intervention (appr. 2 months)
Change from Baseline in Hospital Anxiety and Depression Scale (HADS) depression score at follow-up | Baseline, 3-month follow-up
Change from Baseline in the Quality of Life Scale (QOLS) at the end of intervention (after 5th session) | Baseline, end of intervention (appr. 2 months)
Change from Baseline in the Quality of Life Scale (QOLS) at follow-up | Baseline, 3-month follow-up
Change from Baseline in the European Quality of Life-5 dimensions scale (EQ-5D) at the end of intervention (after 5th session) | Baseline, end of intervention (appr. 2 months)
Change from Baseline in the European Quality of Life-5 dimensions scale (EQ-5D) at follow-up | Baseline, 3-month follow-up

OTHER OUTCOMES:
Change from Baseline in the Self-efficacy-scale (general subscale: GSE) at the end of intervention (after 5th session) | Baseline, end of intervention (appr. 2 months)
Change from Baseline in the Self-efficacy-scale (general subscale: GSE) at follow-up | Baseline, 3-month follow-up
Change from Baseline in the Self-efficacy-scale (social subscale: SSE) at the end of intervention (after 5th session) | Baseline, end of intervention (appr. 2 months)
Change from Baseline in the Self-efficacy-scale (social subscale: SSE) at follow-up | Baseline, 3-month follow-up
Change from Baseline in the Thought control questionnaire (TCQ) at the end of intervention (after 5th session) | Baseline, end of intervention (appr. 2 months)
Change from Baseline in the Thought control questionnaire (TCQ) at follow-up | Baseline, 3-month follow-up
Change from Baseline in the Thought control ability questionnaire (TCAQ) at the end of intervention (after 5th session) | Baseline, end of intervention (appr. 2 months)
Change from Baseline in the Thought control ability questionnaire (TCAQ) at follow-up | Baseline, 3-month follow-up
Change from Baseline in the Behavioural inhibition system and behavioural activation system (BIS/BAS), BAS scale, at the end of intervention (after 5th session) | Baseline, end of intervention (appr. 2 months)
Change from Baseline in the Behavioural inhibition system and behavioural activation system (BIS/BAS), BAS scale, at follow-up | Baseline, 3-month follow-up
Change from Baseline in the Behavioural inhibition system and behavioural activation system (BIS/BAS), BIS scale, at the end of intervention (after 5th session) | Baseline, end of intervention (appr. 2 months)
Change from Baseline in the Behavioural inhibition system and behavioural activation system (BIS/BAS), BIS scale, at follow-up | Baseline, 3-months follow-up
Change from Baseline in health service resource use as measured with a Resource Use Questionnaire | Baseline, 3-months follow-up
Change from before to after scan in the Profile of Mood States (POMS) | Before and after each scanning session (appr. 2 months: session 1: week 1; session 2: week 2; session 3: week 3; session 4: week 4; session 5: week 8)
  Measure to address any imminent changes in mood state.
Relation between upregulation ability of target areas (as obtained by functional MRI analysis) and perceived self control | Integrating imaging and psychometric data across the intervention period (appr. 2 months)
  Analysis of the relationship between scores on the self-efficacy scales, thought control questionnaire (TCQ), thought control ability questionnaire (TCAQ) and the behavioural inhibition system and behavioural activation system (BIS/BAS) scales and fMRI data.

CONTACTS AND LOCATIONS:
Overall Officials: David E Linden, MD, Principal Investigator — Cardiff University
Locations (2):
- United Kingdom (2):
  - CUBRIC, Cardiff, Wales
  - School of Medicine, Cardiff University, Cardiff, Wales

REFERENCES:
- [Background] Johnston SJ, Boehm SG, Healy D, Goebel R, Linden DE. Neurofeedback: A promising tool for the self-regulation of emotion networks. Neuroimage. 2010 Jan 1;49(1):1066-72. doi: 10.1016/j.neuroimage.2009.07.056. Epub 2009 Jul 29. PMID 19646532
- [Background] Johnston S, Linden DE, Healy D, Goebel R, Habes I, Boehm SG. Upregulation of emotion areas through neurofeedback with a focus on positive mood. Cogn Affect Behav Neurosci. 2011 Mar;11(1):44-51. doi: 10.3758/s13415-010-0010-1. PMID 21264651
- [Derived] Fovet T, Jardri R, Linden D. Current Issues in the Use of fMRI-Based Neurofeedback to Relieve Psychiatric Symptoms. Curr Pharm Des. 2015;21(23):3384-94. doi: 10.2174/1381612821666150619092540. PMID 26088117